CLINICAL TRIAL: NCT06631092
Title: An Open-label, Phase I/II Multicenter Clinical Trial of NECVAX-NEO1 as add-on to First-line Neoadjuvant Anti-PD-1 Monoclonal Antibody Therapy in Patients With Triple-negative Breast Cancer
Brief Title: Personalised Neoantigen-targeting Cancer Vaccine NECVAX-NEO1 in Neoadjuvant Triple-negative Breast Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NEC Bio B.V (Industry)
Collaborators: NEC Bio Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NECVAX-NEO1-05-DE; 2024-512520-11-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-02; First posted 2024-10-08 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2024-10

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Vaccines, DNA

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NECVAX-NEO1 (Experimental): Personalised neoantigen-targeting oral DNA cancer vaccine
  Interventions: Biological: Oral DNA Vaccine

INTERVENTIONS:
Biological: Oral DNA Vaccine — Bacteria-based orally administered personalised neoantigen-targeting cancer vaccine

SUMMARY:
Phase I/II, multicenter, open-label, single-arm trial in triple-negative breast cancer patients under first-line neoadjuvant therapy with approved standard of care anti-PD-1 monoclonal antibody (PD-1 inhibitor), epirubicin/cyclophosphamide chemotherapy, and nab-paclitaxel therapy. NECVAX-NEO1 treatment in addition to standard of care anti-PD1 monoclonal antibody therapy can be prolonged after breast cancer surgery for another 24 weeks, according to the investigator's decision taking into consideration the study patient's health status.

DETAILED DESCRIPTION:
Phase I/II, multicenter, open-label, single-arm trial in triple-negative breast cancer patients under first-line neoadjuvant therapy with approved standard of care anti-PD-1 monoclonal antibody (PD-1 inhibitor), epirubicin/cyclophosphamide chemotherapy, and nab-paclitaxel therapy. Optionally, NECVAX-NEO1 treatment in addition to standard of care anti-PD1 monoclonal antibody therapy can be prolonged after breast cancer surgery for another 24 weeks, according to the investigator's decision taking into consideration the study patient's health status.

Personalized NECVAX-NEO1 constructs containing an eukaryotic expression plasmid encoding a series of selected neoantigen epitopes will be manufactured for administration as a patient-specific investigational medicinal product (IMP). The IMP will be administered and as an add-on therapy to the standard of care PD-1 inhibitor therapy.

The trial will consist of mainly:

* A Screening and Induction period of up to 12 weeks, including the neoantigen selection and manufacturing phase, and first-line treatment with PD-1 inhibitor therapy with epirubicin 90 mg/m2/cyclophosphamide 600 mg/m2 every 3 weeks combined with pembrolizumab 200 mg as standard of care treatment,
* A Treatment period of up to 12 weeks with prime and booster administrations of NECVAX-NEO1 in addition to continuation of PD-1 inhibitor pembrolizumab 200 mg every 3 weeks and nab-paclitaxel 125 mg/m2 once a week for 12 weeks up to planned tumor surgery,
* An optional prolongation of booster administration of NECVAX-NEO1 in addition to continuation of PD-1 inhibitor up to 24 weeks, and
* A Follow-up period of 4 weeks, with an End of Treatment (EoT) visit at Week 16 or at Week 40 (in case of the optional treatment prolongation).
* A long-term safety follow-up period (observation period) after EoT for up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients able to understand and follow instructions during the trial.
2. Patients able and willing to give written informed consent, signed and dated.
3. Female and male patients.
4. Patients aged at least 18 years old at the time of ICF signature.
5. cT2-4 N0 or any N-positive (stage II-III) triple-negative breast cancer patients diagnosed as candidates for neoadjuvant anti-PD1 monoclonal antibody and anthracycline/taxane based chemotherapy
6. Patients with tumor accessible for biopsy and surgery and showing at least 30% of tumoral cells on the biopsy.
7. Patients with adequate bone marrow function at Screening, confirmed at Baseline, including:

   1. ANC ≥ 1.5 × 109/L; patients with documented benign cyclical neutropenia are eligible if white blood cell count is ≥ 1.5 × 109/L, with ANC ≥ 1.0 × 109/L, leukocytes ≥ 4.0 × 109/L, and lymphocytes ≥ 0.6 × 109/L;
   2. platelets ≥ 100 × 109/L;
   3. hemoglobin ≥ 9 g/dL (may have been transfused);
8. International Normalized Ratio (INR) < 1.5×Upper Limit of Normal (ULN); patients treated with vitamin K antagonist are eligible if INR < 3.
9. Patients with adequate hepatic function at Screening, confirmed at Baseline, defined by

   1. total bilirubin level ≤1.5×ULN; patients with documented Gilbert disease are allowed if total bilirubin ≤3×ULN;
   2. aspartate aminotransferase (AST) level ≤2.5×ULN, and alanine aminotransferase (ALT) level ≤2.5×ULN, or, for patients with documented metastatic disease to the liver, AST and ALT levels ≤5×ULN.
10. Patients with adequate renal function at Screening, confirmed at Baseline, defined by eGFR ≥ 30 mL/min using 2021 CKD-EPI creatinine equation.
11. Patients must be able to undergo MRI/Ultrasound imaging procedures for tumor follow-up.
12. Patients with Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
13. Life expectancy of at least 12 months according to the Investigator's judgement.

Exclusion Criteria:

Medical and surgical history, and diseases

1. Patients with a history of any disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that, based on the Investigator's judgement, provides a reasonable suspicion of a disease or condition that contraindicates the use of the IMP or that might affect the interpretation of the trial results or render the patient at high risk for treatment complications.
2. Patients with CTCAE v 5.0 Grade 3 or higher not having resolved to Grade 1 within 6 weeks before Baseline.
3. Patients with any significant co-morbidity which, according to the Investigator's judgement, makes patient compliance to trial conditions unlikely.
4. Patients with previous malignant disease (other than the tumor disease for this trial) within the last five (5) years (except adequately treated non-melanoma skin cancers and carcinoma in situ of skin, bladder, cervix, colon/rectum, breast, or prostate) unless a complete remission without further recurrence was achieved at least two (2) years prior to Screening, and the patient is deemed to have been cured with no additional therapy required or anticipated to be required.
5. Patients who underwent prior organ transplantation, including allogeneic stem cell transplantation.
6. Patients with congenital or any other immunodeficiency syndromes, or any active autoimmune disease that might deteriorate when receiving an immunostimulatory agent, except for:

   a. Patients with vitiligo, psoriasis, alopecia not requiring immunosuppressive treatment, are eligible.

   b. Administration of steroids through a route known to result in a minimal systemic exposure (topical, intranasal, intro-ocular, or inhalation), is acceptable.
7. Patients with history of uncontrolled intercurrent illness, including but not limited to uncontrolled hypertension (high blood pressure defined as BPD>=140 mmHg or BPS >=90 mmHg despite of combination therapy with diuretic/CCB/ACE or ARB).
8. Patients with a known prior hypersensitivity or contraindications to any of the IMPs or any component in its formulations or any other drug scheduled or likely to be given during the trial, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v5.0 Grade ≥ 3).
9. Patients with severe acute or chronic medical conditions, including

   1. Immune colitis
   2. Inflammatory bowel disease
   3. History of severe vomiting or diarrhea not having resolved to Grade 1 at Baseline
   4. Immune pneumonitis
   5. Pulmonary fibrosis
   6. Psychiatric conditions including recent (within the last year) or active suicidal ideation or behavior
   7. Laboratory abnormalities that may increase the risk associated with trial participation or trial treatment administration or may interfere with the interpretation of trial results and, in the judgement of the Investigator, would make the patient inappropriate for entry into this trial.
10. Patients with a history of small intestine resection surgery or other major gastrointestinal surgery
11. Patients with active infection requiring systemic therapy with antibiotics (at both Screening and Baseline).
12. Patients with a known history of human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome or multi-drug resistant gram-negative bacteria.
13. Patients with hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at Screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody Screening test positive).
14. Patients with increased anesthesiological risk (e.g. known or predicted difficult airway) if general anesthetic is required .
15. Patients with increased bleeding risk (e.g. coagulopathies) and patients on anticoagulants.
16. Women who are pregnant or breastfeeding, or women of childbearing potential (defined as any woman who is not surgically sterile with a hysterectomy and/or bilateral oophorectomy or ≥ 12 months of amenorrhea and at least 50 years of age) not willing to use highly effective methods of birth control. Highly effective birth control is defined as follows:

    1. combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation 1: • oral

       • intravaginal

       • transdermal
    2. progestogen-only hormonal contraception associated with inhibition of ovulation 1: • oral

       • injectable
       * implantable 2
    3. intrauterine device (IUD) 2
    4. intrauterine hormone-releasing system (IUS) 2
    5. bilateral tubal occlusion 2
    6. vasectomised partner 2,3
    7. sexual abstinence 4

NOTES:

1. Hormonal contraception may be susceptible to interaction with the IMP, which may reduce the efficacy of the contraception method (see section 4.3)
2. Contraception methods that in the context of this guidance are considered to have low user dependency.
3. Vasectomised partner is a highly effective birth control method provided that partner is the sole sexual partner of the WOCBP trial participant and that the vasectomised partner has received medical assessment of the surgical success.
4. In the context of this guidance sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject.

Males of child-bearing potential are to use a highly effective method of birth control to avoid pregnancy with any partner during the study and until the end of the Follow-up period (EoT) or 30 calendar days after the last dose of IMP.

17. Patients with a known history of drug/substance abuse.

Prior and concomitant medication

18. Patients who received any live vaccines within 30 days prior to trial treatment.

19. Patients participating Treatment in any other clinical trial within 30 days before Screening.

20. Patients receiving any other treatment that, in the opinion of the Investigator, might interfere with the trial

21. Patients with a current drug or substance abuse.

22. Patients with chronic concurrent therapy within 2 weeks before the trial treatment or expected therapy during the trial treatment period with:

1. Corticosteroids (except systemic corticosteroids up to 10 mg prednisolone or equivalent daily dose).
2. Immunosuppressive agents.
3. Antibiotics. Any other anticancer therapy or concurrent anticancer treatment except the neoadjuvant chemotherapy / anti-PD1 checkpoint inhibitor standard of care background therapy as per study protocol.

Other 23. Patients unable to understand the Protocol requirements, instructions and trial-related restrictions, the nature, scope, and possible consequences of the trial.

24. Patients who are unlikely to comply with the Protocol requirements, instructions and trial-related restrictions, e.g., uncooperative attitude, inability to return for follow-up visits, and improbability of completing the trial.

25. Patients with legal incapacity or limited legal capacity. 26. Patients with any condition which results in an undue risk for the patient during the trial participation according to the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | Up to 36 weeks plus 24 months
  AEs listed including system organ class, preferred term, severity, causality and other possibly relevant information. Frequency tables (including both patient and event counts) by System Organ Class (SOC) and preferred term (in number and percentage)
Serious Adverse Events | Up to 36 weeks plus 24 months
  SAEs listed including system organ class, preferred term, severity, causality and other possibly relevant information. Frequency tables (including both patient and event counts) by System Organ Class (SOC) and preferred term (in number and percentage)
Change from Baseline in Laboratory Parameters | Up to 36 weeks plus 24 months
  Laboratory defined units
Change from Baseline in Electrocardiograms | Up to 36 weeks plus 24 months
  ECG QT interval

SECONDARY OUTCOMES:
Antitumor activity | Up to 36 weeks
  Changes in ctDNA
Event-free survival | Up to 36 weeks plus 24 months
  Time from first dose of NECVAX-NEO1 to any of the following events: progression of disease that precludes surgery, local or distant recurrence, or death due to any cause up to the end of the safety follow-up at 24 months
Invasive disease-free survival | Up to 36 weeks plus 24 months
  Time from first dose of NECVAX-NEO1 until local or distant recurrence or death due to any cause up to the end of the safety follow-up at 24 month
Residual cancer burden | At week 12
  RCB index
Pathological complete response | At week 12
  Absence of residual invasive cancer

OTHER OUTCOMES:
Tumor immune biomarker | Up to week 12
  Number intratumoral T-cells
Overall survival (OS) | Up to 36 weeks plus 24 months
  Time from first NECVAX-NEO1 administration to death up to the end of the safety follow-up at 24 months
Intestinal microbiome | Up to week 36
  Percentage of bacteria species

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - University Clinic Erlangen, Erlangen
  - National Center for Tumor Diseases Heidelberg, Heidelberg